CLINICAL TRIAL: NCT02167971
Title: Evaluation of Repetitive Transcranial Magnetic Stimulation on the Cognitive Rehabilitation After Traumatic Diffuse Axonal Injury.
Brief Title: Brain Stimulation for Traumatic Brain Injury
Acronym: TMS/DAI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Iuri Santana Neville Ribeiro, iurineville, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USP-01
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Traumatic Brain Injury; Diffuse Axonal Injury
Keywords: traumatic brain injury; diffuse axonal injury; repetitive transcranial magnetic stimulation; neuromodulation; cognitive rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Diffuse Axonal Injury | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Coil (Experimental): The patients assigned to this group will undergo repetitive Transcranial Magnetic Stimulation over 10 sessions (each one with 2,000 pulses) on left dorsolateral prefrontal cortex.
  Interventions: Other: Active Coil
- Sham (Sham Comparator): The patients assigned to this group will undergo 10 sessions of rTMS but with an inactive coil, which will not generate electromagnetic pulses.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Active Coil — The patients will undergo 10 sessions (2,000 pulses each, lasting 20 minutes) of repetitive transcranial magnetic stimulation over the left dorsolateral prefrontal cortex with the following parameters: 10Hz, 50 trains (40 pulses on each train), biphasic wave, 25 seconds between the trains.
  Arms: Active Coil
Other: Sham — The patients assigned to this group will undergo 10 sessions of rTMS but with an inactive coil, which will not generate electromagnetic pulses.
  Arms: Sham

SUMMARY:
The purpose of this study is to determine whether repetitive Transcranial Magnetic Stimulation (rTMS) is effective in the cognitive rehabilitation of patients with diffuse axonal injury(DAI) after Traumatic Brain Injury(TBI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of traumatic brain injury.
* Between one to two years after traumatic brain injuri
* Must be able to sign the Informed Consent Form

Exclusion Criteria:

* Drug addiction
* Uncontrolled epilepsy
* Extensive Cranial vault defects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement on Attentional processes measured by cognitive evaluation (Trail Making Test parts A and B; Stroop Test - Victoria Version; Symbol Digit Test) | One week and three months after rTMS.

SECONDARY OUTCOMES:
Evidence of improvement on Executive Function processes measured by cognitive evaluation. | one week and 3 months.
Evidence of improvement on Motor Coordination measured by cognitive evaluation. | one week and three months.
Changes in cortical excitability measured by single and paired-pulse TMS | one week and three months.

CONTACTS AND LOCATIONS:
Overall Officials: Wellingson S Paiva, MD, Study Chair — University of Sao Paulo; Iuri N Ribeiro, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinics Hospital - University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Rodrigues PA, Zaninotto AL, Ventresca HM, Neville IS, Hayashi CY, Brunoni AR, de Paula Guirado VM, Teixeira MJ, Paiva WS. The Effects of Repetitive Transcranial Magnetic Stimulation on Anxiety in Patients With Moderate to Severe Traumatic Brain Injury: A Post-hoc Analysis of a Randomized Clinical Trial. Front Neurol. 2020 Dec 4;11:564940. doi: 10.3389/fneur.2020.564940. eCollection 2020. PMID 33343483
- [Derived] Neville IS, Zaninotto AL, Hayashi CY, Rodrigues PA, Galhardoni R, Ciampi de Andrade D, Brunoni AR, Amorim RLO, Teixeira MJ, Paiva WS. Repetitive TMS does not improve cognition in patients with TBI: A randomized double-blind trial. Neurology. 2019 Jul 9;93(2):e190-e199. doi: 10.1212/WNL.0000000000007748. Epub 2019 Jun 7. PMID 31175209
- [Derived] Neville IS, Hayashi CY, El Hajj SA, Zaninotto AL, Sabino JP, Sousa LM Jr, Nagumo MM, Brunoni AR, Shieh BD, Amorim RL, Teixeira MJ, Paiva WS. Repetitive Transcranial Magnetic Stimulation (rTMS) for the cognitive rehabilitation of traumatic brain injury (TBI) victims: study protocol for a randomized controlled trial. Trials. 2015 Oct 5;16:440. doi: 10.1186/s13063-015-0944-2. PMID 26438108